CLINICAL TRIAL: NCT06633952
Title: Accelerating Cognitive Gains From Digital Meditation With Noninvasive Brain Stimulation: A Pilot Study in MCI
Brief Title: Accelerating Cognitive Gains From Digital Inverventions With Noninvasive Brain Stimulation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AG080528; R61AG080528 (NIH)
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Aging; MCI
Keywords: healthy aging; cognitive decline; prevention; brain stimulation; attention; memory
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- MediTrain (Experimental)
  Interventions: Device: MediTrain; Device: noninvasive neurostimulation device; Device: wrist worn multi-sensor watches
- Worder (Experimental)
  Interventions: Device: Worder; Device: noninvasive neurostimulation device; Device: wrist worn multi-sensor watches

INTERVENTIONS:
Device: MediTrain — MediTrain is a tablet-based, meditation-inspired, cognitive training game aimed at improving self-regulation of internal attention and distractions. It was developed in collaboration with meditation thought-leader Jack Kornfield, and Zynga, a world-class video game company. It was created to make benefits of concentrative meditation more easily accessible to anyone, including complete novices. This is achieved by creating a game that yields quantifiable and attainable goals, provides feedback, and includes an adaptive algorithm to gradually increase difficulty as users improve.
  Arms: MediTrain
Device: Worder — Worder was designed to enhance visual motor and visual spatial skills in individuals of all ages and cognitive abilities. Visual processing is required for all cognitive abilities that involve vision including attention, working memory, and task management. Worder's goal is to improve cognitive function more broadly by developing this critical skill underlying multiple abilities.
  Arms: Worder
Device: noninvasive neurostimulation device — A noninvasive neurostimulation device will be used to deliver theta frequency stimulation or sham stimulation to the frontal part of the brain.
Device: wrist worn multi-sensor watches — Stress and sleep data will be recorded at home throughout the intervention using FDA-approved wrist worn multi-sensor watches.

SUMMARY:
The overall goal of this project is to collect pilot feasibility and early efficacy data showing improvements in cognition and wellbeing in adults with mild cognitive impairment (MCI) through a combination treatment of non-invasive brain stimulation (transcranial alternating current stimulation (tACS)) and a one of two digital cognitive interventions.

ELIGIBILITY:
comfortably ambulatory healthy physical condition normal or corrected to normal visual auditory acuity fluency in spoken English Between 60-85 years old No neurological or psychiatric disorders No substance abuse Not taking anti-depressants Not taking anti-anxiety medication No history of seizures No color blindness No glaucoma No macular degeneration No amblyopia (lazy eye) No strabismus (cross eyed) Aneurysm clip(s) No Cardiac pacemaker No Implanted cardioverter defibrillator (ICD) No Electronic implant or device No Magnetically-activated implant or device No Neurostimulation system No Spinal cord stimulator No Internal electrodes or wires No Bone growth/bone fusion stimulator No Cochlear, otologic, or other ear implant No Insulin or other infusion pump No Implanted drug infusion device No type of prosthesis (eye, penile, etc.) No Heart valve prosthesis No Eyelid spring or wire No Artificial or prosthetic limb No Metallic stent, filter, or coil No Shunt (spinal or intraventricular) No Vascular access port and/or catheter No Radiation seeds or implants No Swan-Ganz or thermodilution catheter No Medication patch (Nicotine, Nitroglycerine) No metallic fragment or metallic foreign body in/on the body that can not be removed No Wire mesh implant No Tissue expander (e.g., breast) No Surgical staples, clips, or metallic sutures No Joint replacement (hip, knee, etc.) No Bone/joint pin, screw, nail, wire, plate, etc. No IUD, diaphragm, or pessary No Dentures or partial plates that can not be removed No Tattoo or permanent makeup No Body piercing jewelry No Claustrophobia

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-09-13 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Mean change on the Continuous Performance Task (CPT) over time | baseline and immediate follow-up
  The CPT is a 23-minute task, where participants are instructed to respond to target stimuli (squares at the top of the screen) and withhold responses to non-target stimuli (squares at the bottom of the screen). Performance will be quantified as: (1) mean reaction times, (2) standard deviation of reaction times (RTV), and (3) d-prime (comparing correct target detections or 'hits' to incorrect non-target detections or 'false alarms').

SECONDARY OUTCOMES:
Mean change in Telomere length | baseline and immediate follow-up
  200 mL of blood will be collected from each participant before and after the intervention. Blood will be centrifuged for whole blood cell acquisition and stored at -80 °C for subsequent batch testing. Telomere length (T/S ratio) will be quantified in peripheral blood mononuclear cells.
Mean change on a distracted attention task over time | baseline and immediate follow-up
  Mean performance on a distracted attention task will be compared pre and post intervention. Divided attention performance will be assessed using the Filter Task that places simultaneous demands on perceptual discrimination abilities and distraction filtering.
Mean Change in Frontal Theta Power over time | baseline and immediate follow-up
  Based on previous studies of meditation training and our preliminary data, we predict that MediTrain will lead to significantly enhanced midline frontal theta power during the TOVA in MCI as compared to OA. Beyond most prior studies, by collecting structural MRI data, we will be able to source-localize any observed changes in midline frontal theta.
Mean change in resting state networks over time | baseline and immediate follow-up
  We also expect MediTrain will augment intrinsic Default Mode Network (DMN) connectivity, both functionally (measured with resting fMRI111,112) and structurally (measured with DTI-based connectomes). This is hypothesized based on the known association between the DMN

OTHER OUTCOMES:
Mean change on the Adaptive Cognitive Evaluation (ACE) over time | baseline and immediate follow-up
  The ACE is a mobile cognitive assessment tool, which includes a battery of cognitive control tests for rapid tests of cognition. The sub-tests (or 'modules') in ACE are adapted from standardized tasks to rapidly assess various aspects of cognition, including attention, memory, and multitasking. We will assess response time, accuracy, and response time variability in each case, with faster/more accurate/less variable performance being indicative of improved cognitive control, meditation, and frontal theta power.
Mean change in continuous recordings of sleep and stress metrics. | baseline and immediate follow-up
  We will assess time spent in NonREM stages 1 (N1), 2 (N2) and 3 (N3) sleep and REM sleep (RS), latency to sleep onset (SOL), and wake after sleep onset (WASO). We will also assess delta power during sleep stages and wake; and overall sleep maintenance (SM) and sleep efficiency (SE). Diminished time spent in SOL and WASO, increased time N2, N3 and REM sleep, increased delta during NonREM sleep are each signs of improved sleep. Increases in SM and SE indicated improved, more stable sleep patterns. We will measure continuous pulse rate, heart rate variability, respiration, electrodermal activity , and peripheral skin temperature. Reduced amplitude can be indicative of reduced stress over time.
Mean change in Change in Mnemonic Discrimination over time | baseline and immediate follow-up
  Mnemonic discrimination task tests recognition memory for common objects, as reported in scores on a scale of the Lure Discrimination Index ranging from 0.00 to 1.00 where higher values show better performance.
Mean change in Task-based Cortical Functional Connectivity | baseline and immediate follow-up
  Changes in Task-based Cortical Functional Connectivity Associated With Training-induced Changes in Mnemonic Discrimination will be measured. functional MRI data will be analyzed in terms of beta-series correlations between co-active cortical regions of interest and compared between treatment arms and timepoints.
Mean Change on Everyday Cognition Scale (ECog) | baseline and immediate follow-up
  The Everyday Cognition Scale (ECog) measures the ability to perform everyday tasks that demand memory, language, visuospatial abilities, planning, organization, and divided attention. The ECog consists of a global and domain scores for each of the previously described categories, and is scored as follows: 1= better or no change compared to 10 years earlier, 2= questionable/occasionally worse compared to 10 years earlier, 3= consistently a little worse compared to 10 years earlier, 4= consistently much worse compared to 10 years earlier. Thus, the lower the overall score is on this measure at both the global and domain score level, the better one is performing with respect to their cognition.
Mean Change on SF-36 (overall health) | baseline and immediate follow-up
  SF-36 (overall health) The general health and well-being (SF-36) score assesses participant health. The SF-36 score ranges from 0 to 100. The higher the overall score is on this measure, the better one is performing with respect to their health and well-being.
Mean Change on Perceived Stress Scale | baseline and immediate follow-up
  Perceived Stress Scale A survey that measures the degree to which situations in one's life are perceived as stressful. Scores range from 0 to 40 with higher scores representing more perceived stress. We will report change in means over time.

CONTACTS AND LOCATIONS:
Overall Officials: David Ziegler, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No